CLINICAL TRIAL: NCT01789580
Title: Moderators of Online Gambling, How Effective? Experimental, Controlled and Randomized Study.
Brief Title: MOD&JEU: Moderators of Online Gambling, How Effective?
Acronym: MOD&JEU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC12_0153
Record Dates: First submitted 2013-02-06; First posted 2013-02-12 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Online Gambling
Keywords: Experimental study, moderators, online gambling,; problem gambling prevention

ARMS (5):
- Control group (No Intervention): The participants play on their preferred online gambling site (experimental gambling session) without gambling moderator.
- Bonus group (Experimental): The participants play on their preferred online gambling site (experimental gambling session) with the first gambling moderator sudied : bonus (with different modalities of the moderator).
  Interventions: Other: Gambling moderator
- Auto-exclusion group (Experimental): The participants play on their preferred online gambling site (experimental gambling session) with the first gambling moderator sudied : auto-exclusion.
  Interventions: Other: Gambling moderator
- Auto- limitation group (Experimental): The participants play on their preferred online gambling site (experimental gambling session) with the first gambling moderator sudied : auto- limitation(with different modalities of the moderator).
  Interventions: Other: Gambling moderator
- Information group (Experimental): The participants play on their preferred online gambling site (experimental gambling session) with the first gambling moderator sudied : information (with different modalities of the moderator).
  Interventions: Other: Gambling moderator

INTERVENTIONS:
Other: Gambling moderator
  Other Names: The intervention consists in leaving the participants play on their; preferred online gambling site.; The participant will be randomly assigned to an experimental condition; (i.e. the implementation of the gambling session with the presence of the; moderator studied) or to the control condition (i.e. with no moderator present).
  Arms: Auto- limitation group; Auto-exclusion group; Bonus group; Information group

SUMMARY:
Prevalence of problem gambling is estimated about 1-3% of the general adult population. This percentage increases to 5% when talking about online gambling. In France, the market for online gambling was recently opened up to competition and regulation (May 2010), including poker and sports/horse races betting, but excluding for the moment casino games. Recent international studies show that legalizing online gambling led to an increase of practices, including problem gambling.

In France, the law stipulates the establishment of moderators of online gambling, to prevent excessive gambling practices. The Regulatory Authority of Online Games (ARJEL) guarantees the implementation of these moderators. However, no evaluation of the effectiveness of these moderators is planned.

Therefore the investigators propose to conduct an experimental study about online gambling. The objective will be to evaluate the effectiveness of four kinds of moderators, some already legislated, but not evaluated, and others offered by the investigators team. Proposals for amending legislation will be made according the results of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* French people, living around Nantes
* Giving their consent for access to their gambling account
* User of a gambling site approved by the ARJEL, with an active account
* Regular gambler (gambling at least once a week, since at least 3 months)

Exclusion Criteria:

* Age under 18 and over 65
* Excessive gamblers (CPGI > 8) or gambler seeking treatment
* Protected persons (pregnant women, being under protection measures)
* Overindebtedness
* Psychiatric or cognitive major dysfunctions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 485 (Estimated)
Dates: Start 2013-02; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of studied moderators | 2 month
  Impact on money wagered and time spent gambling during the experimental gambling session (measured at the end of the gambling session +/- 15 days after +/- 2 months after, depending on the tested moderator)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc VENISSE, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Caillon J, Grall-Bronnec M, Saillard A, Leboucher J, Pere M, Challet-Bouju G. Impact of Warning Pop-Up Messages on the Gambling Behavior, Craving, and Cognitions of Online Gamblers: A Randomized Controlled Trial. Front Psychiatry. 2021 Jul 23;12:711431. doi: 10.3389/fpsyt.2021.711431. eCollection 2021. PMID 34366941
- [Derived] Challet-Bouju G, Grall-Bronnec M, Saillard A, Leboucher J, Donnio Y, Pere M, Caillon J. Impact of Wagering Inducements on the Gambling Behaviors, Cognitions, and Emotions of Online Gamblers: A Randomized Controlled Study. Front Psychiatry. 2020 Nov 17;11:593789. doi: 10.3389/fpsyt.2020.593789. eCollection 2020. PMID 33312142
- [Derived] Caillon J, Grall-Bronnec M, Hardouin JB, Venisse JL, Challet-Bouju G. Online gambling's moderators: how effective? Study protocol for a randomized controlled trial. BMC Public Health. 2015 May 30;15:519. doi: 10.1186/s12889-015-1846-7. PMID 26024922